CLINICAL TRIAL: NCT00003968
Title: Phase II Study of Bryostatin-1 in Metastatic Renal Cell Carcinoma(Summary Last Modified 8/1999)
Brief Title: Bryostatin 1 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02303; FCCC-99012; NCI-T99-0002; CDR0000067169 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2004-01

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — bryostatin 1

ARMS (1):
- Arm I (Experimental): Patients receive bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment continues every 4 weeks in the absence of unacceptable toxicity or disease progresssion.
  Interventions: Drug: bryostatin 1

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
Phase II trial to study the effectiveness of bryostatin 1 in treating patients who have metastatic kidney cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate to bryostatin 1 in patients with advanced renal cell carcinoma.

II. Assess the toxicities of this treatment regimen in this patient population. III. Determine the time to disease progression in patients receiving this treatment regimen.

IV. Determine the overall survival of this patient population treated with this regimen.

OUTLINE:

Patients receive bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment continues every 4 weeks in the absence of unacceptable toxicity or disease progresssion.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma
* Bidimensionally measurable disease
* Clear evidence of progression if only site of measurable disease is within previous radiation port
* Previously irradiated brain metastases allowed, if not life threatening, symptoms controlled for 3 months, and not requiring corticosteroids

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-1
* Life expectancy: Greater than 3 months
* WBC at least 3,000/mm3
* Platelet count at least 100,00/mm3
* Bilirubin no greater than 1.5 mg/dL
* Creatinine no greater than 2.0 mg/dL OR creatinine clearance greater than 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for 3 months after study
* No active bacterial or viral infection
* No serious underlying medical condition that would interfere with compliance
* No other malignancy within the past 5 years except basal cell carcinoma of the skin
* No dementia or altered mental status that would prevent informed consent

PRIOR CONCURRENT THERAPY:

* No more than 1 prior therapy with biologic response modifiers
* No prior chemotherapy for advanced disease
* No other concurrent chemotherapy
* No concurrent steriods (except topical use)
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* At least 4 weeks since major surgery (including nephrectomy)
* No other concurrent experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1999-06; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S. Balzer-Haas, MD, Study Chair — Fox Chase Cancer Center
Locations (17):
- United States (17):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Medical Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania